CLINICAL TRIAL: NCT05883683
Title: Precision Medicine for Advanced or Recurrent Colorectal Cancer Directed by High-throughput Sequencing and Tumor Organoids Model
Brief Title: Molecular Study and Precision Medicine for Colorectal Cancer
Acronym: MSPM
Status: Not yet recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zheng Wang, MD/PhD, Study chair, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: CIT-CoPT-R01
Record Dates: First submitted 2022-07-12; First posted 2023-06-01 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Advanced Colorectal Carcinoma; Recurrent Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour samples will be collected for molecular characterization and organoids establishment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Colorectal Cancer: Colorectal cancer patients with advanced or recurrent tumors
  Interventions: Other: Molecular Profiling & drug testing in tumor organoids and PDXs

INTERVENTIONS:
Other: Molecular Profiling & drug testing in tumor organoids and PDXs — Molecular profiling of native tumor will be performed and analyzed by using a self-designed panel. Tumor organoids will be cultured from fresh tumor tissues and patient-derived xenografts model will be established using the tumor organoids. Drugs will be tested in the two models. And the recommendation will be communicated to the clinicians.

SUMMARY:
Researchers collect specimens from advanced or recurrent colorectal cancer (CRC) patients to conduct molecular profiling and establish tumor organoids (PDOs)/ patient-derived xenografts (PDXs). The aim of this study is to identify clinical actionable targets and predict in vivo response of the tumor to targeted drugs by using PDOs/ PDXs. And the above-mentioned studies will provide the patients with potential personalized cancer treatment options.

DETAILED DESCRIPTION:
Patient-derived organoid is a model that can recapitulate the histology and behavior of the cancer from which it is derived, and is increasingly used as a tool for drug development in pre-clinical settings. Clinical treatment option of colorectal cancer now is quite limited. By molecular profiling, clinical actionable alterations may be identified. And according to the genomic investigation results, we can find the matched targeted drugs, following further testing in the organoids and PDXs. This will provide an opportunity to guide the precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age 18 to 75 years old
* Patients with a documented (histologically- or cytologically-proven) advanced or recurrent colorectal cancer
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status =< 1 and a life expectancy of at least 3 months
* Patients, both male and female, who are either not of childbearing potential or who agree to use a medically effective method of contraception during the study and for 3 months after the last dose of study drug.
* Patients with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol.

Exclusion Criteria:

* Patients with any other life-threatening illness, significant organ system dysfunction, or clinically significant laboratory abnormality, which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluation of the safety of the study drug
* Patients with abnormal coagulation function, bleeding tendency, or receiving thrombolytic or anticoagulant therapy
* Patients with any other serious/active/uncontrolled infection, any infection requiring parenteral antibiotics, or unexplained fever > 38ºC within 2 weeks prior to first study drug administration.
* Patients with a history of human immunodeficiency virus (HIV) or any other immunodeficiency disease.
* Patients who are currently using certain drugs that are not permitted
* Patients with a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies
* Patients with the inability, in the opinion of the Investigator, to comply with the protocol requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced or recurrent colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Identification of effective drugs or drug combinations | up to 3 years
  Viability of organoid is measured using CellTiter-Glo by quantifying ATP, which indicates the presence of metabolically active cells.

SECONDARY OUTCOMES:
Comparison of clinical actionable alterations identified in native tumor and organoids. | Up to 3 years
  Genomic gene mutation numbers are identified using the Next-Generation Sequencing (NGS).
Correlation between organoid and PDX drug sensitivities | Up to 3 years
  Size of the tumor is measured to reflect the drug response.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Wang, MD/PhD, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pauli C, Hopkins BD, Prandi D, Shaw R, Fedrizzi T, Sboner A, Sailer V, Augello M, Puca L, Rosati R, McNary TJ, Churakova Y, Cheung C, Triscott J, Pisapia D, Rao R, Mosquera JM, Robinson B, Faltas BM, Emerling BE, Gadi VK, Bernard B, Elemento O, Beltran H, Demichelis F, Kemp CJ, Grandori C, Cantley LC, Rubin MA. Personalized In Vitro and In Vivo Cancer Models to Guide Precision Medicine. Cancer Discov. 2017 May;7(5):462-477. doi: 10.1158/2159-8290.CD-16-1154. Epub 2017 Mar 22. PMID 28331002